CLINICAL TRIAL: NCT02518685
Title: Endoscopic Treatment for Weight Reduction in Patients With Obesity Using the TransPyloric Shuttle® System: A Multicenter, Prospective, Randomized, Double-Blind, Sham-Controlled, Parallel-Design Study
Brief Title: ENDObesity® II Study: TransPyloric Shuttle® System for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BaroNova, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DTC006
Record Dates: First submitted 2015-08-06; First posted 2015-08-10 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Device; Non-surgical; Endoscopic; TransPyloric Shuttle; TPS
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TransPyloric Shuttle (TPS) (Experimental): TransPyloric Shuttle plus Lifestyle Counseling
  Interventions: Device: TransPyloric Shuttle; Behavioral: Lifestyle Counseling
- Control (Sham Comparator): Sham procedure plus Lifestyle Counseling
  Interventions: Device: Sham procedure; Behavioral: Lifestyle Counseling

INTERVENTIONS:
Device: TransPyloric Shuttle
  Other Names: TPS
  Arms: TransPyloric Shuttle (TPS)
Device: Sham procedure
  Arms: Control
Behavioral: Lifestyle Counseling — The goal of lifestyle modification counseling is to promote adherence to a reduced calorie diet, increased physical activity and to recommend behavioral modification strategies.

SUMMARY:
The purpose of this clinical research trial is to study safety and effectiveness of the TransPyloric Shuttle System (TPSS) for weight reduction in patients who are considered medically obese.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 22 to 60
* A BMI between 30.0 to 40.0 kg/m2, inclusive. Subjects with a BMI of 30.0 kg/m2 to 34.9 kg/m2 are required to have one or more obesity-related comorbidities
* History of obesity for at least 2 years, with history of failure of medically or commercially supervised weight loss program
* < 5% change in body weight for at least 3 months
* Negative pregnancy test, agree to be on birth control for the duration of participation
* Informed consent
* Willing and able to comply with study procedures

Exclusion Criteria:

* Pregnancy or nursing
* Hormonal or genetic cause for obesity
* Prior history of any GI surgery or endoscopic intervention
* Chronic use of medications likely to contribute to weight gain or prevent weight loss
* Gastric or duodenal ulcers
* Positive for H. pylori
* History of severe dyspepsia
* GI tract motility disorders
* History of inflammatory disease of GI tract, coeliac disease, pancreatitis, portal hypertension, cirrhosis, and/or varices
* Diabetes treated with insulin
* HbA1c >7.5%
* Uncontrolled thyroid and adrenal gland disease or uncontrolled hypertension
* History of certain cardiac events
* Localized or systemic infection
* Anemia
* History of asthma likely to require systemic steroid therapy
* Autoimmune connective tissue disorders or immunocompromised
* History of malignancy except non-melanoma skin cancer
* Continuous use of ulcerogenic medication
* On anticoagulation or antiplatelet therapy
* Use of weight-loss medication
* In other weight-loss program
* Unable to take proton pump inhibitor
* Abnormal laboratory values or EKG
* Inability to walk at least 0.8 kilometers per day
* Planned surgical procedure that can impact the conduct of the study
* Known allergy to any component materials in the TPSS
* Smoker or user of nicotine product
* Substance abuse
* Severe, uncontrolled psychiatric illness
* Recent inpatient psychiatric treatment
* Moderate depression
* Bulimia nervosa or binge eating disorder
* Participation in another clinical study
* Employee or family member of Sponsor or study staff
* Have any endoscopic exclusion criteria

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 302 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard I Rothstein, MD, Principal Investigator — Dartmouth Geisel School of Medicine
Locations (9):
- United States (9):
  - HonorHealth Bariatric Center, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - University of Miami, Miami, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Stony Brook Medicine, Stony Brook, New York
  - MidSouth Bariatrics, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TransPyloric Shuttle (TPS) | Control
Started (Subjects randomized) | 213 | 89
Safety Cohort (Ten subjects did not receive TPS) | 203 (Randomized to and successfully received TPS (171) + Open-Label TPS-treated Subjects (32)) | 89
Randomized Cohort | 181 | 89
Enrolled | 213 (Includes 171 Successful device deployments, 10 unsuccessful delivery attempts and 32 Open-Label) | 89
Per Protocol Analysis | 168 (Three TPS-treated subjects were inadvertently unblinded, excluding them from efficacy analyses.) | 89
Completed (Completed 12-Month Visit) | 164 (Randomized Completers (139) plus Open-Label Completers (25)) | 79
Not Completed | 49 | 10
Not completed — Adverse Event | 29 | 1
Not completed — Withdrawal by Subject | 10 | 3
Not completed — relocation, study fatigue | 7 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TransPyloric Shuttle (TPS) | Control | Total
Number analyzed (Participants) | 181 | 89 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 181 | 89 | 270
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (8.9) | 43.9 (8.5) | 43.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 83 | 252
  Male | 12 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 12 | 40
  Not Hispanic or Latino | 153 | 77 | 230
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 32 | 13 | 45
  White | 131 | 65 | 196
  More than one race | 13 | 6 | 19
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 181 | 89 | 270

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Total Body Weight Loss (% TBL) Between the TPS and the Control Group
Description: The mean percent Total Body Weight Loss (% TBL) is the percentage weight change at 12 Months from Baseline
Time Frame: 12 Months
Measure: Least Squares Mean (Standard Error); unit: % Total Body Weight Loss
Groups:
- TransPyloric Shuttle (TPS): TransPyloric Shuttle plus lifestyle counseling
  TransPyloric Shuttle
  lifestyle counseling
- Control: Sham procedure plus lifestyle counseling.
  lifestyle counseling
  Sham procedure
Arm/Group | TransPyloric Shuttle (TPS) | Control
Number analyzed (Participants) | 168 | 89
% Total Body Weight Loss | 9.5 (0.65) | 2.8 (0.87)
Statistical Analysis 1: Comparison: TransPyloric Shuttle (TPS) vs Control; Test type: Superiority; p < 0.0001, multiple imputations; Least-Square Mean Difference = 6.7, 95% CI 2-sided [4.54 to 8.81]

2. Primary Outcome: Proportion of TPS-treated Subjects With Weight Loss ≥ 5% TBL
Description: The proportion of subjects in the TPS group with ≥ 5% TBL is compared to a performance target of 50%
Time Frame: 12 months
Population: Per Protocol Population; received TPS Device
Measure: Count of Participants; unit: Participants
Arm/Group | TransPyloric Shuttle (TPS)
Number analyzed (Participants) | 168
Participants | 112
Statistical Analysis 1: Comparison: TransPyloric Shuttle (TPS); Test type: Superiority — Statistical success criterion for achieving the performance standard of (≥ 50%) of proportion of TPS subjects who have 5% or more TBL at the 12-Month Follow-up; p < 0.0001, Wilson's Midpoint Estimate; Proportion of Subjects = 66.8, 95% CI 2-sided [59.3 to 74.3]

ADVERSE EVENTS:
Time Frame: 12 months
Description: The TPS, SAE population includes all subjects successful deliveries plus 10 subjects with attempted deliveries.
  The TPS, AE population includes successful deliveries where the TPS remained for up to one year
Arm/Group | TransPyloric Shuttle (TPS) | Control
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/89
Serious Adverse Events (participants affected / at risk) | 10/213 | 1/89
Other Adverse Events (participants affected / at risk) | 203/203 | 87/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TransPyloric Shuttle (TPS) (N=213) | Control (N=89)
esophageal rupture (Gastrointestinal disorders) | 1 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — due to esophageal rupture in same patient
upper abdominal pain (Gastrointestinal disorders) | 1 | 0
gastric ulcer (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 0
device intolerance (General disorders) | 1 | 0
gastric obstruction (Gastrointestinal disorders) | 1 | 0
cerebrovascular accident (Nervous system disorders) | 0 | 1 — not device or procedure related
cholelithiasis (Hepatobiliary disorders) | 3 | 0 — not device or procedure related
divericularitis (Gastrointestinal disorders) | 1 | 0 — not device or procedure related
meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — not device or procedure related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TransPyloric Shuttle (TPS) (N=203) | Control (N=89)
nausea (Gastrointestinal disorders) | 131 | 35
abdominal pain upper (Gastrointestinal disorders) | 128 | 37
vomiting (Gastrointestinal disorders) | 126 | 14
dyspepsia (Gastrointestinal disorders) | 113 | 31
diarrhea (Gastrointestinal disorders) | 105 | 29
abdominal distension (Gastrointestinal disorders) | 77 | 17
gastroesophageal reflux (Gastrointestinal disorders) | 72 | 23
eructation (Gastrointestinal disorders) | 67 | 9
constipation (Gastrointestinal disorders) | 47 | 8
gastritis, erosive (Gastrointestinal disorders) | 29 | 3
gastric mucosa erythema (Gastrointestinal disorders) | 25 | 3
gastric ulcer (Gastrointestinal disorders) | 21 | 0
abdominal pain (Gastrointestinal disorders) | 17 | 1
abdominal pain lower (Gastrointestinal disorders) | 15 | 3
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 75 | 44
nasopharyngitis (Infections and infestations) | 12 | 11
esophageal mucosal injury (Injury, poisoning and procedural complications) | 18 | 8 — endoscopic observations during procedure
pyrexia (General disorders) | 12 | 3
pain (General disorders) | 11 | 3
headache (Nervous system disorders) | 16 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02518685/Prot_SAP_000.pdf